CLINICAL TRIAL: NCT05328973
Title: Intraoperative Aromatherapy Versus Placebo for Port-a-Cath Placement Under Monitored Anesthesia Care. A Randomized Controlled Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-0994; NCI-2022-03112 (Other: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2022-04-05; First posted 2022-04-14 (Actual); Results first posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Cancer Pain
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ELEQUIL (Other): Aromatherapy will be provided using a lavender-peppermint patch called an Aromatab.
  Interventions: Other: ELEQUIL

INTERVENTIONS:
Other: ELEQUIL — patch placed on skin
  Other Names: Aromatabs

SUMMARY:
This is a prospective, controlled, randomized trial. Primary objective is to compare the time to readiness for discharge (minutes) from Post-Anesthesia Care Unit (PACU) after Port-a-Cath placement surgery between patients who are randomized to receive intraoperative aromatherapy versus placebo. 70 Eligible subjects will be identified from within the patient population of the study site. There will be no advertisements for study subjects.

DETAILED DESCRIPTION:
Primary Objective:

To compare the time to readiness for discharge (minutes) from Post-Anesthesia Care Unit (PACU) after Port-a-Cath placement surgery between patients who are randomized to receive intraoperative aromatherapy versus placebo.

Secondary Objective:

To evaluate the following secondary outcomes:

* Anxiety score (HADS) in preoperative holding area
* Midazolam use intraoperatively (mg)
* Itraoperative opioid use (morphine equivalents)
* Intraoperative anti-emetic use
* Time to first occurrence of postoperative nausea or vomiting (PONV) in PACU
* Rate and intensity of PONV in PACU
* Antiemetic use in PACU
* Opioid use in PACU (morphine equivalents)
* Pain intensity in PACU (0-10 numerical rating scale)
* Patient satisfaction in PACU

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old)
* Port-a-Cath placement under Monitored Anesthesia Care
* Signed informed consent

Exclusion Criteria:

* Patients undergoing other surgical procedures during Port-a-Cath placement (including explantation of a Port-a-Cath or other previous vascular access device)
* Patients requiring general anesthesia or those not eligible for MAC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Bailard, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Bailard N, Cukierman DS, Guerra-Londono JJ, Brown E, Hagberg C, Sauer A, Cata JP. Use of a Combination Lavender/Peppermint Aromatherapy Patch During Port Catheter Placement Under Monitored Anesthesia Care Does Not Reduce Time to Discharge Readiness: A Randomized Controlled Trial. J Integr Complement Med. 2024 Sep;30(9):840-847. doi: 10.1089/jicm.2023.0416. Epub 2024 Mar 19. PMID 38502819
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled 70 patients between May 2022 and March 2023. Eligible subjects were identified from within the patient population of the study site by members of the research team.
Groups:
- Elequis Aromatab (Lavander/Pepermint): Elequis Aromatab was placed next to patient's pillow
- Placebo: Placebo tab was placed next to patient's pillow
Period: Overall Study
Arm/Group | Elequis Aromatab (Lavander/Pepermint) | Placebo
Started | 35 | 35
Completed | 35 | 34
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elequis Aromatab (Lavander/Pepermint) | Placebo | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.4 (13.225) | 52.886 (15.212) | 52.64 (14.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 26 | 54
  Male | 7 | 9 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Count of Participants; unit: Participants] — Subject were staged according to their Body Mass Index in the two categories below.
  Participants
    <=25 | 13 | 13 | 26
    >25 | 22 | 22 | 44
ASA [Count of Participants; unit: Participants] — American Society of Anesthesiologists Physical Status Classification ranges from 1 to 6, where 1 is for a normal healthy patient, and 6 for a Brain-dead patient whose organs are being harvested. During this study, patients with a classification 2 & 3 qualified and enrolled.
  Participants
    2 | 3 | 0 | 3
    3 | 32 | 35 | 67
Charlson Score [Count of Participants; unit: Participants] — CCI score ranged from 0 to 11. The scores were categorized into the following groups: 0, 1-2, 3-4, and >=5. A higher score means high comorbid disease increasing anesthesia risk.
  Participants
    0 | 1 | 3 | 4
    1 to 2 | 8 | 11 | 19
    3 to 4 | 15 | 6 | 21
    >=5 | 11 | 15 | 26

OUTCOME MEASURES:

1. Primary Outcome: To Compare the Time to Readiness for Discharge From PACU (Minutes) After Port-a-Cath Placement Surgery Between Patients Who Are Randomized to Receive Intraoperative Aromatherapy Versus Placebo
Description: It measures the time to readiness for discharge from PACU (minutes) from PACU arrival to PACU discharge ready
Time Frame: from "PACU arrival" to "PACU discharge ready", 1.5 hrs in average
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Elequis Aromatab (Lavander/Pepermint) | Placebo
Number analyzed (Participants) | 35 | 34
Minutes | 82.057 (15.376) | 89.382 (21.25)

2. Secondary Outcome: Anxiety Score (HADS) in Preoperative Holding Area
Description: The Hospital Anxiety and Depression Scale (HADS) is a self-report questionnaire that measures anxiety and depression. The HADS has 14 items, divided into two subscales of seven items each, and each item is scored on a 4-point Likert scale ranging from 0-3. Scores are interpreted as follows: 0-7: Normal 8-10: Borderline 11-21: Abnormal
Time Frame: From "In preop" to "Preop end" per EMR. 1hr in average
Measure: Count of Participants; unit: Participants
Arm/Group | Elequis Aromatab (Lavander/Pepermint) | Placebo
Number analyzed (Participants) | 35 | 34
Participants
  Abnormal | 1 | 2
  Borderline | 3 | 3
  Normal | 31 | 29

3. Secondary Outcome: Midazolam Use Intraoperatively (mg)
Description: The use on intravenous Midazolam in mg as per Anesthesia record.
Time Frame: From "Anesthesia Start" to "Anesthesia End". 1hr in average
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Elequis Aromatab (Lavander/Pepermint) | Placebo
Number analyzed (Participants) | 35 | 34
mg | 3.63 (1.28) | 3.6 (1.5)

4. Secondary Outcome: Opioid Use Intraoperatively (in MEDD)
Description: The use on intravenous opioids as per Anesthesia record, converted to MEDD (morphine milligram equivalent daily dose)
Time Frame: From "Anesthesia Start" to "Anesthesia End". 1hr in average
Measure: Mean (Standard Deviation); unit: MEDD
Arm/Group | Elequis Aromatab (Lavander/Pepermint) | Placebo
Number analyzed (Participants) | 35 | 34
MEDD | 2.59 (1.05) | 2.91 (1.5)

5. Secondary Outcome: Intraoperative Anti-emetic Use
Description: The use on intravenous Ondansetron in mg as per Anesthesia record.
Time Frame: From "Anesthesia Start" to "Anesthesia End". 1hr in average
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Elequis Aromatab (Lavander/Pepermint) | Placebo
Number analyzed (Participants) | 35 | 34
mg | 4 (0.97) | 3.41 (1.43)

6. Secondary Outcome: Number of Participants With Postoperative Nausea or Vomiting (PONV) in PACU
Description: Measured in assessments done at 1, 15, 30 minutes from PACU start. Patients were asked for nausea or vomiting.
Time Frame: From "PACU Start" to "PACU Discharge", 1.5 hr in average
Measure: Count of Participants; unit: Participants
Arm/Group | Elequis Aromatab (Lavander/Pepermint) | Placebo
Number analyzed (Participants) | 35 | 34
Participants | 0 | 1

7. Secondary Outcome: Rate and Intensity of PONV in PACU
Description: Measured using the Verbal Numeric Rating Scale (0: no nausea and 10 worst nausea ever), patients were asked how would they rate their PONV.
Time Frame: From "PACU Start" to "PACU Discharge", 1.5 hr in average
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elequis Aromatab (Lavander/Pepermint) | Placebo
Number analyzed (Participants) | 35 | 34
score on a scale | 0 (0) | 0.0118 (0.0686)

8. Secondary Outcome: Anti-emetic Use in PACU
Description: Number of Patients given antiemetic medication in PACU
Time Frame: From "PACU Start" to "PACU Discharge", 1.5 hr in average
Measure: Count of Participants; unit: Participants
Arm/Group | Elequis Aromatab (Lavander/Pepermint) | Placebo
Number analyzed (Participants) | 35 | 24
Participants | 0 | 1

9. Secondary Outcome: Opioid Use in PACU
Description: Number of Patients given opioids in PACU
Time Frame: From "PACU Start" to "PACU Discharge", 1.5 hr in average
Measure: Count of Participants; unit: Participants
Arm/Group | Elequis Aromatab (Lavander/Pepermint) | Placebo
Number analyzed (Participants) | 35 | 34
Participants | 2 | 3

10. Secondary Outcome: Pain Intensity in PACU (0-10 Numerical Rating Scale)
Description: Pain intensity reported by the patients during their stay in PACU, using the the numerical rating scale (NRS) 0 to 10, whereas 0 means no pain, and 10 means the worst possible pain.
Time Frame: From "PACU Start" to "PACU Discharge", 1.5 hr in average
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elequis Aromatab (Lavander/Pepermint) | Placebo
Number analyzed (Participants) | 35 | 34
score on a scale | 0.3257 (1.0371) | 0.5429 (1.0661)

11. Secondary Outcome: Patient Satisfaction in PACU
Description: Rating the experience in PACU by the patients using the Likert Scale
Time Frame: From "PACU Start" to "PACU Discharge", 1.5 hr in average
Measure: Count of Participants; unit: Participants
Arm/Group | Elequis Aromatab (Lavander/Pepermint) | Placebo
Number analyzed (Participants) | 35 | 34
Participants
  Unknown | 0 | 0
  Somewhat satisfied | 0 | 2
  Very much satisfied | 35 | 32

ADVERSE EVENTS:
Time Frame: From "Anesthesia Start" to "PACU Discharge", approximately 3 hours.
Description: Number of patients who reported Adverse Events or were observed by health providers
Arm/Group | Elequis Aromatab (Lavander/Pepermint) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 1/35 | 3/34
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elequis Aromatab (Lavander/Pepermint) (N=35) | Placebo (N=34)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Transient Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT05328973/Prot_SAP_000.pdf